CLINICAL TRIAL: NCT07133711
Title: Impact of Noninvasive Ventilation Weaning Protocol on Outcome of Patients With Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: Noninvasive Ventilation Weaning Protocol in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Waleed Gamal Elddin Khaleel, Assistant professor of chest diseases, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WGEK-NIV-Weaning-Trial
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Noninvasive ventilation; Weaning
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: Each participant is assigned to only one of the three intervention groups (gradual pressure support decrement, gradual time spent on noninvasive per day decrement, abrupt withdrawal of noninvasive ventilatory support) for the entire duration of the weaning period.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the interventions, participants and clinical staff managing the weaning will not be blinded to group assignment. However, outcome assessors [the physician adjudicating weaning success based on predefined criteria] and data analysts will be blinded to group allocation throughout the outcome assessment and analysis phases
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gradual PS Decrement (Experimental): ): pressure support will be reduced by 2-4 cm H2O every 6-8 h with vitals and blood gas monitoring till IPAP of <8 cm of H2O and EPAP of <4 cm of H2O is attained, after which NIV will be completely withdrawn
  Interventions: Device: Noninvasive ventilation
- Gradual Time Decrement (Experimental): the duration of NIV will be reduced to 16 h on the day of randomization (day 0), then reduced to 12 h on day 1 (including 6-8 h of overnight use), 6-8 h of overnight use on day 2, and complete withdrawal on day 3.
  Interventions: Device: Noninvasive ventilation
- Abrupt Withdrawal (Active Comparator): patients will be immediately withdrawn from NIV and monitored on spontaneous breathing.
  Interventions: Device: Noninvasive ventilation

INTERVENTIONS:
Device: Noninvasive ventilation — Weaning from noninvasive ventilation for patients with acute exacerbation of COPD

SUMMARY:
Noninvasive ventilation (NIV) has revolutionized the management of patients with acute exacerbation of chronic obstructive pulmonary disease (AECOPD) with hypercapnic respiratory failure (HcRF). NIV use has been shown to reduce the need for endotracheal intubation, hospital and intensive care unit (ICU) length of stay, and mortality.

Multiple studies have been conducted on weaning strategies among patients requiring invasive mechanical ventilation. As a result of these studies, definite criteria and protocols have been laid down for weaning from invasive mechanical ventilation. However, no such data are available for the withdrawal of NIV.

Evidence-based reviews suggest that protocols to manage the weaning and liberation of subjects from Mechanical Ventilation could reduce the time that subjects spend receiving mechanical ventilation. However, no such data about protocolized withdrawal of NIV are available.

DETAILED DESCRIPTION:
A study to compare protocolized weaning from non-invasive ventilation using three potential strategies of weaning from NIV

* Stepwise reduction of duration of NIV use,
* Stepwise reduction in pressure support of NIV, and
* Immediate withdrawal of NIV. Among patients with Acute respiratory failure due to acute exacerbation of COPD.

ELIGIBILITY:
Inclusion Criteria:

* All COPD patients admitted in the respiratory ICU with acute Hypercapnic Respiratory Failure who will be managed with Noninvasive Ventilation without the need for invasive mechanical ventilation will be eligible for inclusion in the study.

Exclusion Criteria:

* Age: less than 18 years,
* End organ failure as cardiac/ Liver/ Renal,
* Patients on home NIV and
* Those who required NIV for respiratory failure due to diseases other than COPD were not considered for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Successful weaning | 48 hours
  The primary objective of the study is to compare the rate of successful withdrawal of NIV among the three groups.

CONTACTS AND LOCATIONS:
Overall Officials: waleed gamal elddin, ass. prof, Principal Investigator — Assiut University
Locations (1):
- Assiut University hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davidson AC, Banham S, Elliott M, Kennedy D, Gelder C, Glossop A, Church AC, Creagh-Brown B, Dodd JW, Felton T, Foex B, Mansfield L, McDonnell L, Parker R, Patterson CM, Sovani M, Thomas L; BTS Standards of Care Committee Member, British Thoracic Society/Intensive Care Society Acute Hypercapnic Respiratory Failure Guideline Development Group, On behalf of the British Thoracic Society Standards of Care Committee. BTS/ICS guideline for the ventilatory management of acute hypercapnic respiratory failure in adults. Thorax. 2016 Apr;71 Suppl 2:ii1-35. doi: 10.1136/thoraxjnl-2015-208209. No abstract available. PMID 26976648
- [Background] Lun CT, Chan VL, Leung WS, Cheung AP, Cheng SL, Tsui MS, Chu CM. A pilot randomized study comparing two methods of non-invasive ventilation withdrawal after acute respiratory failure in chronic obstructive pulmonary disease. Respirology. 2013 Jul;18(5):814-9. doi: 10.1111/resp.12080. PMID 23490403
- [Background] Brochard L, Rauss A, Benito S, Conti G, Mancebo J, Rekik N, Gasparetto A, Lemaire F. Comparison of three methods of gradual withdrawal from ventilatory support during weaning from mechanical ventilation. Am J Respir Crit Care Med. 1994 Oct;150(4):896-903. doi: 10.1164/ajrccm.150.4.7921460.